CLINICAL TRIAL: NCT00005066
Title: A Phase II Trial of O6-Benzylguanine (NSC 637037) and BCNU (Carmustine) in Patients With Advanced Soft Tissue Sarcoma
Brief Title: O6-benzylguanine and Carmustine in Treating Patients With Recurrent, Metastatic, or Locally Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10227; UCCRC-10227; UCCRC-T99-0088; NCI-T99-0088
Record Dates: First submitted 2000-04-06; First posted 2004-04-12 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Sarcoma
Keywords: recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — O(6)-benzylguanine; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): O6-BG as an intravenous infusion (through your vein) over 1 hour followed 1 hour later by BCNU intravenously over 15 minutes. chemotherapy every 6 weeks.
  Interventions: Drug: O6-benzylguanine; Drug: carmustine

INTERVENTIONS:
Drug: O6-benzylguanine
Drug: carmustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining O6-benzylguanine and carmustine in treating patients who have recurrent, metastatic, or locally advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate of patients with recurrent, metastatic, or locally advanced soft tissue sarcoma treated with O6-benzylguanine and carmustine. II. Determine the toxicity of this regimen in this patient population. III. Determine the duration of response, time to progression, and survival of these patients treated with this regimen.

OUTLINE: Patients receive O6-benzylguanine IV over 1 hour followed 1 hour later by carmustine IV over 15 minutes. Treatment continues every 6 weeks for a minimum of 2 courses in the absence of unacceptable toxicity or disease progression. Patients with progressive disease are followed every 6 months until death. Patients without progressive disease are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 12-35 patients will be accrued for this study within 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed recurrent, metastatic, or locally advanced soft tissue sarcoma considered incurable by surgery or radiotherapy Bidimensionally measurable disease At least 1 cm x 1 cm, with clearly defined margins on CT scan, X-ray, or physical examination Located outside of radiation port or evidence of progression within radiation port No CNS disease only No uncontrolled symptomatic brain metastases regardless of other disease sites

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal unless due to Gilbert's syndrome SGOT or SGPT no greater than 2 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Pulmonary: DLCO at least 80% predicted Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other concurrent significant underlying medical or psychiatric illness (e.g., active infection) that would preclude study treatment or exceptionally increase risk of toxicities No other prior malignancy within the past 5 years except curatively treated nonmelanoma skin cancer, carcinoma in situ of the cervix, or superficial bladder cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for metastatic disease At least 4 weeks since prior neoadjuvant and/or adjuvant chemotherapy No other concurrent chemotherapy No concurrent investigational antineoplastic drugs Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 3 weeks since prior radiotherapy and recovered No concurrent radiotherapy to any lesion Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2000-06; Primary Completion 2001-09 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Disease response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Walter M. Stadler, MD, FACP, Study Chair — University of Chicago
Locations (10):
- United States (10):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Division of Hematology/Oncology, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana